CLINICAL TRIAL: NCT00916786
Title: Pharmacogenetic Studies on Attention Deficit Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 200812153M
Record Dates: First submitted 2009-06-08; First posted 2009-06-10 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: Attention-deficit/hyperactivity disorder; pharmacogenetics; molecular genetics; medication response
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The subjects will receive blood withdrawal. The blood sample will be used for establishing lymphoblastoid cell lines, which will be used for molecular genetic experiments.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- OROS-methylphenidate: The patients will be randomly assigned to two treatment groups, the OROS-methylphenidate group (n=80) and the atomoxetine group (n=80), respectively.
- Atomoxetine group: The patients will be randomly assigned to two treatment groups, the OROS-methylphenidate group (n=80) and the atomoxetine group (n=80), respectively.
- Control group: Healthy controls matching for the distribution of age and sex of the case groups

SUMMARY:
The ultimate goal of this study is to find the association between specific polymorphism of candidate genes and medication response in attention deficit hyperactivity disorder (ADHD) patients. These results will lead the investigators' team: (1) to resolve controversies over inconsistent findings in previous pharmacogenetic studies; (2) to study the medication effect on the neuropsychological functions that are useful candidate endophenotypes for ADHD; (3) to delineate the nature and the effect of gene-gene interaction in the drug response of ADHD patients.

DETAILED DESCRIPTION:
Background: The science of pharmacogenetics seeks to identify patterns of genetic variation that will direct individually tailored treatment regimens and enhance long-term adherence. Attention deficit hyperactivity disorder (ADHD), characterized by inattention, hyperactivity and impulsivity, is an early onset, highly heritable, clinically heterogeneous, long-term impairing disorder with tremendous impact on individuals, families, and societies. It affects 5-10% of school-aged children worldwide (7.5% in Taiwan) and 2-4% of adults. Although the efficacy of medications for ADHD is well demonstrated in clinical trials, substantial numbers of patients fail to remain on therapy, and there is tremendous variability in tolerability and treatment acceptance. An understanding of genetic predictors of ADHD medication response is likely to influence future clinical treatments, inform research on treatment-resistant ADHD patients, and identify patients at increased risk for significant treatment related adverse events. Although interest in ADHD pharmacogenetics is encouraging, conflicting results in previous studies may reflect genetic heterogeneity and differences in phenotype, and medication response in ADHD children likely results from the combined effects of several potential genes. In addition, the categorical measure of treatment effects and retrospective study design may not have been sensitive enough to pick up statistically significant differences in treatment response based on genotype. Further prospective studies including quantitative measures of medication response are warranted.

Specific Aims:

1. to assess the specific genetic moderators of methylphenidate and atomoxetine response using repeated outcome measurements;
2. to examine the association between genetic polymorphisms and medication effects on the neuropsychological functions;
3. to identify the gene-gene interactions in pharmacogenetics for ADHD. Subjects and Methods: We will recruit 160 drug-naïve ADHD patients and 80 matched normal controls, aged 7-18. The patients will be randomly assigned to two treatment groups, the OROS-methylphenidate group (n=80) and the atomoxetine group (n=80), respectively. After complete assessment at baseline and administration of either OROs-methylphenidate or atomoxetine, patients with ADHD will be reassessed at Week 2, 4, 8, 12, 16, and 24 mainly for vital signs, behavioral symptoms, and psychosocial functions evaluations using the SNAP-IV, YSR, CBCL, CGI-ADHD-S, CGI-ADHD-I, SAICA, and Family APGAR-C. Neuropsychological tests, including CPT, Time Perception Tasks, and CANTAB, will be performed at Week 4 and 16. The DNA will be collected, and the candidate genes (DAT1, DRD4, DRD5, SLC6A2, and SLC6A4) hypothesized to influence medication effects or individual risks for ADHD will be genotyped.

Anticipated Results: We anticipate that this study will delineate the pharmacogenetics for ADHD by determining the association between medication response and genetic variants in a Taiwanese sample. The findings of different approaches to identify the effects of genotypes on the drug response in this study should help us to extend our understanding of the genetic basis of ADHD. Development of individualized medication regimens based on patient genetic variability might lead to optimized symptom reduction, improved tolerability, and concomitant improvements in patient adherence. Conversely, patients with increased genetic risk for treatment failure or significant adverse effects could be spared exposure to certain compounds that are of unlikely benefit. Pharmacogenetics also has a potential role in the development of new compounds for ADHD therapy. The use of genetic screening in dosing will provide a model for future drug development, in which outcome variability is assessed in genetic subgroups and not merely on the basis of treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in this study only if they meet all of the following criteria:

1. Patients will be outpatients who are between 7 and 18 years of age.
2. Patients must have ADHD that meet the Diagnostic and Statistical Manual of Mental disorders, 4th edition (DSM-IV) disease diagnostic criteria assessed by the investigator's clinical evaluation, as well as confirmed by the Chinese version of the Schedule for Affective Disorders and Schizophrenia for School-Age Children-Epidemiological Version (K-SADS-E).
3. Patients must have a Clinical Global Impressions-ADHD-Severity (CGI-ADHD-S) score > 4 at Visit 1.
4. Patients must be psychotropic medication-naïve. Patients will be considered to be medication-naïve if they have never received medications specifically to treat ADHD.
5. Patients must have laboratory results, including serum chemistries, hematology, and urine analysis showing no significant abnormalities and no clinical information that should preclude a patient's participation at study entry. A patient with a significant abnormal laboratory result mat enter the study if, after appropriate medical evaluation, the result dose not indicate a serious medical condition that in the investigator's judgment would preclude participation.
6. Patients and parents (or legal representative) must have a degree of understanding sufficient to be able to communicate suitably with the investigator.
7. Patients must be of normal intelligence in the judgment of the investigator. Normal intelligence is defined as achieving a score of 80 or more when IQ testing is administrated.
8. Patients must have been judged by the investigator to be reliable to keep appointments for clinic visits and all tests, including neuropsychological testing and venipunctures.

Exclusion Criteria:

Patients will be excluded from the study if they meet any of the following criteria:

1. Patients with current or past history of schizophrenia, schizoaffective Disorder, organic psychosis, bipolar I or II disorder, autism, Asperger's disorder, or pervasive developmental disorder. Other comorbid psychiatric disorders are not excluded if the ADHD symptoms are the primary source of impairment for the patient.
2. Patients with a history of any seizure disorder (other than febrile convulsion) or patients who are taking anticonvulsants for seizure control.
3. Patients have been at serious suicidal risk, determined by the investigator.
4. Patients with a history of severe allergies to more than one class of medications or multiple adverse drug reactions.
5. Patients with a history of alcohol or drug abuse within the past 3 months, or who are currently using alcohol, drugs of abuse, or any described or over-the-counter medication in a manner that the investigator considers indicative of abuse.
6. Patients with cardiovascular disease or other conditions that could be aggravated by an increased heart rate or increased blood pressure.
7. Patients who are likely to need psychotropic medications apart from methylphenidate or atomoxetine, including Chinese medicine or health-food supplements that have central nervous system activity.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The sample will consist of 160 drug-naïve ADHD patients and 80 matched normal controls, aged 7-18. The patients will be randomly assigned to two treatment groups, the OROS-methylphenidate group (n=80) and the atomoxetine group (n=80), respectively.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2009-08-01 (Actual); Primary Completion 2012-07-31 (Actual); Study Completion 2012-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chi-Yung Shang, MD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Wu CS, Shang CY, Lin HY, Gau SS. Differential Treatment Effects of Methylphenidate and Atomoxetine on Executive Functions in Children with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2021 Apr;31(3):187-196. doi: 10.1089/cap.2020.0146. PMID 33890819
- [Derived] Chou TL, Chia S, Shang CY, Gau SS. Differential therapeutic effects of 12-week treatment of atomoxetine and methylphenidate on drug-naive children with attention deficit/hyperactivity disorder: A counting Stroop functional MRI study. Eur Neuropsychopharmacol. 2015 Dec;25(12):2300-10. doi: 10.1016/j.euroneuro.2015.08.024. Epub 2015 Sep 8. PMID 26409297
- [Derived] Shang CY, Pan YL, Lin HY, Huang LW, Gau SS. An Open-Label, Randomized Trial of Methylphenidate and Atomoxetine Treatment in Children with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2015 Sep;25(7):566-73. doi: 10.1089/cap.2015.0035. Epub 2015 Jul 29. PMID 26222447